CLINICAL TRIAL: NCT02129504
Title: Comparison of Two Surgical Techniques to Optimize the Treatment of Gingival Recessions Using a Gingival Graft Substitute.
Brief Title: Two Techniques for Root Coverage With a Xenogeneic Collagen Matrix
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Arthur Belem Novaes Jr, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PCM
Record Dates: First submitted 2014-04-29; First posted 2014-05-02 (Estimated); Last update posted 2014-05-02 (Estimated); Status verified 2014-05

CONDITIONS: Gingival Recession
Keywords: root coverage; gingival recession; periodontal surgery
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- coronal advanced technique (Experimental): root coverage with the porcine collagen matrix using the coronal advanced technique (standard technique)
  Interventions: Device: root coverage comparing two techniques
- extended flap technique (Experimental): root coverage with the porcine collagen matrix using the extended flap technique (new surgical technique)
  Interventions: Device: root coverage comparing two techniques

INTERVENTIONS:
Device: root coverage comparing two techniques — The aim of this study was to compare and show the benefits of the extended flap technique (new technique) compared to coronal advanced technique (gold standard technique) both techniques using the porcine collagen matrix for root coverage.
  Other Names: Mucograft; porcine collagen matrix; extended flap technique; coronal advanced flap technique

SUMMARY:
Gingival recessions are often successfully treated by coronally advanced flap technique (CAF) associated with subepithelial connective tissue grafts (SCTG). Currently the xenogeneic collagen matrix (CM) has been used as a substitute for SCTG associated with CAF technique for root coverage. CAF technique was not developed for use with CM and has shown limited results when applied to the CM. The aim of this study was to compare and show the benefits of the extended flap technique (EFT) compared to CAF technique using CM for root coverage.

ELIGIBILITY:
Inclusion Criteria:

* ages 25 to 50 years old
* bilateral gingival recession type Miller class I or II
* with 3 mm in height and less than 3mm of keratinized tissue
* non-molar teeth

Exclusion Criteria:

* diabetics
* pregnant women
* chronic use of medication
* periodontitis

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-09; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Comparing changes for Root coverage measure (in millimeter) from baseline at 3, 6 and 12 months | Change from Baseline at 3, 6 and 12 months
  At the mid-buccal point of the involved tooth, the gingival recession height was measure by the same operator, who was previously calibrated (intra-examiner calibration) using a digital paquimeter.

CONTACTS AND LOCATIONS:
Locations (1):
- School of dentistry of Ribeirão Preto, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Background] McGuire MK, Scheyer ET. Xenogeneic collagen matrix with coronally advanced flap compared to connective tissue with coronally advanced flap for the treatment of dehiscence-type recession defects. J Periodontol. 2010 Aug;81(8):1108-17. doi: 10.1902/jop.2010.090698. PMID 20350159